CLINICAL TRIAL: NCT04956432
Title: A Multicentre, Randomized, Double-blind, Allopurinol Controlled Study to Evaluate the Efficacy and Safety of SHR4640 in Subjects With Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR4640-303
Record Dates: First submitted 2021-07-07; First posted 2021-07-09 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — ruzinurad; Allopurinol

STUDY DESIGN:
Intervention Model Description: To evaluate the efficacy and safety of SHR4640 monotherapy tablets in patients with gout
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): SHR4640+Allopurinol Placebo；once a day, orally, for 52 weeks
  Interventions: Drug: SHR4640
- Treatment group B (Active Comparator): Allopurinol+ SHR4640 Placebo；once a day, orally, for 52 weeks.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: SHR4640 — SHR4640 Dose 1 ,tablets, QD
  Arms: Treatment group A
Drug: Allopurinol — Allopurinol 300mg, tablets, QD
  Arms: Treatment group B

SUMMARY:
This study will assess the serum uric acid lowering effects and safety of SHR4640 compared to Allopurinol in subjects with gout.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who met 1977 or 2015 ACR (American College of Rheumatology) classification of Gout and has a serum acid ≥ 480 μmol/L at screening; 2、18 kg/m2 ≤ Body mass index (BMI) ≤ 35 kg/m2.

Exclusion Criteria:

1. Subject who is pregnant or breastfeeding;
2. Alanine aminotransferase or Aspartate aminotransferase or total bilirubin>1.5 upper normal limit;
3. Subject with a positive test for HLA-B*5801;
4. Estimated glomerular filtration rate (MDRD formula) <60ml/min;
5. HbA1c≥8%;
6. Subject with known hypersensitivity or allergy to SHR4640 and allopurinol, or any component of SHR4640;
7. Subject with kidney stones or suspicion of kidney stones;
8. Subject who has acute gout flares within 2 weeks before randomization;
9. Subject with a history of malignancy within the previous 5 years;
10. Subject with a history of active peptic ulcer within a year;
11. Subject with a history of xanthine urine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a serum uric acid level≤360 μmol/L | Start of Treatment to end of study (approximately 16 weeks)

SECONDARY OUTCOMES:
Percentage change in serum uric acid from baseline at each visit during 16 weeks of treatment | Start of Treatment to end of study (approximately 16 weeks)
Absolute changes in serum uric acid from baseline at each visit during 16 weeks of treatment | Start of Treatment to end of study (approximately 16 weeks)
The proportion of subjects with A serum uric acid level≤ 360 μmol/L at each visit within 16 weeks of treatment | Start of Treatment to end of study (approximately 16 weeks)
Percentage change of serum uric acid from baseline at each visit within 52 weeks of treatment | Start of Treatment to end of study (approximately 52 weeks)
change value of serum uric acid from baseline at each visit within 52 weeks of treatment | Start of Treatment to end of study (approximately 52 weeks)
proportion of subjects with serum uric acid ≤ 360 μmol/L at each visit within 52 weeks of treatment | Start of Treatment to end of study (approximately 52 weeks)
serum uric acid value at each visit within 52 weeks of treatment | Start of Treatment to end of study (approximately 52 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi Hospital, Shanghai JiaoTong University School Of Medicine, Shanghai, Shanghai Municipality, China